CLINICAL TRIAL: NCT04096417
Title: A Phase II, Multicenter, Single-Arm Study of Pemigatinib in Patients With Metastatic or Unresectable Colorectal Cancer Harboring FGFR Alterations
Brief Title: Pemigatinib for the Treatment of Metastatic or Unresectable Colorectal Cancer Harboring FGFR Alterations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-GI-1701; NCI-2019-05877 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1701 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Results first posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-11

CONDITIONS: FGFR1 Gene Amplification; FGFR1 Gene Mutation; FGFR1 Gene Translocation; FGFR2 Gene Amplification; FGFR2 Gene Mutation; FGFR2 Gene Translocation; FGFR3 Gene Amplification; FGFR3 Gene Mutation; FGFR3 Gene Translocation; Metastatic Colorectal Carcinoma; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pemigatinib) (Experimental): Patients receive pemigatinib PO QD on days 1-21. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pemigatinib; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Pemigatinib — Given PO
  Other Names: INCB054828
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well pemigatinib works in treating patients with colorectal cancer with mutations (alterations) in a FGFR gene and that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Pemigatinib may stop the growth of tumor cells by blocking FGFR, which is needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess overall response rate (ORR) of pemigatinib in patients with metastatic or unresectable colorectal cancer harboring activating FGFR alterations.

SECONDARY OBJECTIVES:

I. To assess the clinical benefit rate (complete response + partial response + stable disease) with pemigatinib.

II. To assess progression free survival (PFS) and overall survival (OS) with pemigatinib.

III. Assess changes in patient quality of life (QOL) as measured by the linear analogue self-assessment (LASA) questionnaire.

IV. Assess the frequency and severity of adverse events.

CORRELATIVE RESEARCH OBJECTIVES:

I. To assess plasma pharmacodynamic biomarkers of response and resistance to therapy.

II. To explore any correlation between tissue and blood based biomarkers and clinical outcomes.

OUTLINE:

Patients receive pemigatinib orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Registered to Colorectal and Liquid Biopsy Molecularly Assigned Therapy (COLOMATE) Academic and Community Cancer Research United (ACCRU)-GI-1611 and:

  * COLOMATE Companion Trial Recommendation Form indicates patient qualifies to be screened for a COLOMATE companion trial
  * COLOMATE Companion Trial Recommendation Form date of completion is =< 30 days prior to registration
* Histologically or cytologically confirmed diagnosis of metastatic or unresectable colorectal cancer (mCRC), based on documentation from local or outside review of pathology according to each site?s established institutional procedure
* Documentation of an activating genomic alteration(s) in FGFR1-3 (gain of function mutations, translocations, and amplifications allowed)
* Provide informed written consent
* Patient must have received and progressed on, or be intolerant to, each of the following treatments for mCRC (or have contraindication to these treatments):

  * Fluoropyrimidine
  * Oxaliplatin
  * Irinotecan
  * Anti-VEGF (vascular endothelial growth factor) monoclonal antibody, if eligible for this therapy
  * Anti-EGFR (epidermal growth factor receptor) monoclonal antibody, if eligible for this therapy
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 28 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained =< 28 days prior to registration)
* Total bilirubin =< 1.5x upper limit of normal (ULN), or =< 2.5x ULN if patient has Gilbert syndrome or disease involving the liver (obtained =< 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5x ULN (or =< 5x ULN in presence of suspected liver metastases) (obtained =< 28 days prior to registration)
* Serum phosphate < institutional ULN (obtained =< 28 days prior to registration)
* Serum calcium within institutional normal range, or serum albumin-corrected calcium within institutional normal range (if serum albumin is outside of the institutional normal range) (obtained =< 28 days prior to registration)
* Potassium levels > institutional lower limit of normal (supplementation can be used to correct potassium level during screening) (obtained =< 28 days prior to registration)
* Serum creatinine =< 1.5x ULN, or calculated creatinine clearance > 30 mL/min using the Cockcroft-Gault formula or 24-hours urine collection analysis (obtained =< 28 days prior to registration)
* Corrected QT interval (QTc) by Fridericia?s method (QTcF) assessed by electrocardiogram (ECG) completed =< 28 days prior to registration, and resulted as:

  * QTcF =< 450 msec in men, or
  * QTcF =< 470 msec in women
* Negative serum pregnancy test completed =< 7 days prior to registration, for women of childbearing potential only
* Willing to provide tissue and blood samples for correlative research purposes
* Willing to allow transfer of tissue and blood samples, clinical information, and outcome data collected from this trial for future research

Exclusion Criteria:

* Prior treatment with pemigatinib
* Prior treatment with a selective FGFR inhibitor =< 180 days (6 months) prior to registration
* Known hypersensitivity or severe reaction to an FGFR inhibitor, or to the excipients of pemigatinib (i.e. microcrystalline cellulose, sodium starch glycolate, and magnesium stearate)
* Current evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination
* Treatment with other investigational study drug for any indication for any reason, or receipt of anticancer medications =< 14 days prior to registration
* Major surgery =< 28 days prior to registration
* External beam radiation therapy =< 28 days prior to registration, or palliative radiation for non-central nervous system (CNS) disease =< 14 days prior to registration
* Brain metastases, central nervous system (CNS) metastases, leptomeningeal disease, or spinal cord compression

  * NOTE: Patients who are asymptomatic or previously treated and stable, without evidence of progression for >= 28 days prior to registration are eligible
  * NOTE: Patients taking concomitant corticosteroids and/or anticonvulsants are allowed if patient is on a stable or decreasing dose of such treatment for >= 28 days prior to registration
* History or presence of significant cardiovascular disease or condition including:

  * Uncontrolled angina pectoris (Canadian Cardiovascular Society grade II-IV despite medical therapy)
  * Congestive heart failure (New York Heart Association class III or IV)
  * Uncontrolled arrhythmia requiring therapy. Note: Patients with a pacemaker and well-controlled rhythm for >= 28 days prior to registration are not excluded
  * Any of the following occurring =< 6 months prior to registration: myocardial infarction, angioplasty, cardiac stenting, coronary/peripheral artery bypass graft, cerebrovascular accident or transient ischemic attack
* Failure to adequately recover (i.e. to =< grade 1 [according to Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5] or to pre-treatment baseline) from adverse events (AEs) deemed by the investigator as clinically significant and attributed to prior therapy. Exception: alopecia
* Current use of prohibited medication
* Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers =< 14 days or 5 half-lives (whichever is shorter) prior to registration. Note: topical ketoconazole will be allowed
* History of hypovitaminosis D requiring supraphysiologic doses to replenish the deficiency. Note: patients receiving vitamin D food supplements are allowed
* History and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung; with the exception of calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcification
* Unable or unwilling to swallow pemigatinib and keep a medication diary, or significant gastrointestinal disorder(s) that could interfere with absorption, metabolism or excretion of pemigatinib per the discretion of the investigator
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or men able to father children who have a female partner of childbearing potential, who are unwilling to employ acceptable contraception
* Known history of human immunodeficiency (HIV) infection or positivity on immunoassay confirmed per local standards

  * Note: HIV test is not required for screening, but patients with a known history of HIV infection will be excluded
* Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Other known active malignancy =< 5 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma in situ of the cervix, provided there is no known active disease and no additional therapy for the condition is ongoing or required during the trial period
  * NOTE: anti-estrogen/androgen therapy or bisphosphonates allowed
* Co-morbid systemic illness, other severe concurrent disease, or psychiatric illness/social situation which, in the judgment of the investigator, would make the patient inappropriate for entry into this study, limit compliance with study requirements, or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2025-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen K Ciombor, Principal Investigator — Academic and Community Cancer Research United
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Wheless MC, Zemla TJ, Hubbard JM, Strickler JH, Gbolahan OB, Wilson L, Waechter B, Ou FS, Nixon AB, Bekaii-Saab TS, Ciombor KK. A phase II, multicenter, single-arm study of pemigatinib in patients with metastatic or unresectable colorectal cancer harboring FGFR alterations. Oncologist. 2025 Jun 4;30(6):oyaf069. doi: 10.1093/oncolo/oyaf069. PMID 40515475

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pemigatinib)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 60.5 [36 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Defined as the rate of patients, among evaluable patients, who experience an objective response per RECIST 1.1. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Clopper and Pearson.
Time Frame: 4.4 Months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
proportion of participants | 0.0 [0.0 to 0.232]

2. Secondary Outcome: Clinical Benefit Rate
Description: Clinical Benefit Rate is defined as the number of patients that experience a complete or partial response, or have stable disease, divided by the number of evaluable patients. Analysis of this endpoint will mirror that of the primary objective.
Time Frame: 4.4 Months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
proportion of participants | 0.0 [0.0 to 0.232]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from study entry to the first of either disease progression or death from any cause, where disease progression is determined based on RECIST 1.1 criteria. PFS will be estimated using the Kaplan-Meier method. The median PFS and corresponding 95% confidence interval will be reported. Patients who do not experience disease progression or death while on protocol will be censored at the last disease assessment date.
Time Frame: 4.4 Months
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
Weeks | 9.1 [7.9 to NA] — Not enough events occurred to calculate the upper limit

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from study entry to death from any cause. Will be estimated using the Kaplan-Meier method. The median OS and corresponding 95% confidence interval will be reported.
Time Frame: 29.4 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
Months | 7.9 [3.4 to NA] — Not enough event occurred to calculate the upper limit

5. Secondary Outcome: Quality of Life (QOL) as Measured by the LASA [Item 1: Overall QOL]
Description: Quality of Life (QOL) was measured using item 1: Overall QOL of the Linear Analogue Self-Assessment (LASA) Questionnaire on a 0-10 scale, with 0=as bad as it can be and 10=as good as it can be. The QOL scores was converted to a 100-point scale, with 0=Low QOL and 100=Best QOL. Change from baseline to Week 36 will be calculated by subtracting the baseline scores from the scores at Week 36. Negative change indicates the QOL decrease and positive change indicates the QOL improvement.
Time Frame: 9 Months
Population: All patients that completed and submitted the baseline and week 36 Linear Analogue Self-Assessment.
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 11
score on a scale | -0.1 (1.22)

6. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events will be summarized by frequency and severity using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in the adverse event section of this report. The number of patients evaluated for adverse events is reported below.
Time Frame: 5.4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pemigatinib)
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 5.4 months and mortality was followed for 29.4 months
Arm/Group | Treatment (Pemigatinib)
All-Cause Mortality (participants affected / at risk) | 11/14
Serious Adverse Events (participants affected / at risk) | 6/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pemigatinib) (N=14)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pemigatinib) (N=14)
Anemia (Blood and lymphatic system disorders) | 10 (22)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (16)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (21)
Gait disturbance (General disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (9)
Alkaline phosphatase increased (Investigations) | 9 (17)
Aspartate aminotransferase increased (Investigations) | 8 (15)
Blood bilirubin increased (Investigations) | 5 (7)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 5 (9)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 10 (19)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT04096417/Prot_SAP_000.pdf